CLINICAL TRIAL: NCT01934855
Title: Evaluation of Tumor Motion Management Strategies in Radiotherapy Using 4D-MRI
Brief Title: Tumor Motion Management in Radiotherapy Using 4D-MRI
Status: Completed | Type: Observational
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Other Study IDs: J1370; NA_00085958 (Other: Johns Hopkins Institutional Review Board)
Record Dates: First submitted 2013-08-30; First posted 2013-09-04 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Cancer
Keywords: cancer; radiotherapy; 4D-MRI; 4D-CT; MRI
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The main goal of this research is to characterize patient-specific respiration-induced tumor and surrogate motion to evaluate the accuracy and effectiveness of the surrogate-based motion management strategies currently used in clinics. Specifically, the investigators hypothesize that dynamic MRI (Magnetic Resonance Imaging) obtained over a temporal duration consistent with radiotherapy treatments will provide spatio-temporal information of both the tumor and surrogate, and therefore can serve as a means to assess the quality of the tumor motion tracking with the surrogate. To test this hypothesis, the investigators specifically propose to 1) track and characterize the tumor and surrogate motion with 4D (4 dimensional)-MRI and 2) evaluate surrogate-based motion tracking in a cohort of patients with thoracic tumors.

External and internal surrogate-based strategies commonly used in clinics have not been appropriately validated. With the increasing adaptation of these surrogate methods for motion management, the proposed research addresses these urgent issues in clinical radiotherapy while providing a means to achieve patient-specific motion management.

DETAILED DESCRIPTION:
Respiration-induced patient motion has become a major obstacle for achieving high-precision radiotherapy of cancers especially in the thorax and upper abdomen. As the target is continuously moving, an additional margin has to be added to the clinical target volume to compensate for the uncertainty in the tumor and organ motion, causing toxicity to the normal tissue and limiting the dose delivered to the target. To account for the tumor motion, surrogate tracking methods are commonly used in clinics during radiotherapy. However, the relationship between the surrogate and tumor motion is hard to generalize as it depends on individual patients, tumor location, treatment fractions, and sometimes shows complex patterns or transient, unpredictable changes. Hence, there is an urgent need to better scrutinize the current surrogate-based motion management strategies. Moreover, the most robust motion management strategy for the given patient should be determined in the pre-treatment setting but the investigators currently lack a sufficient tool to provide this information.

4D-CT is typically used to characterize the tumor motion over the course of the radiotherapy. However, 4D-CT is an oversimplified snapshot representation of a single-breathing cycle with low soft tissue contrast while imparting a considerable amount of radiation dose to the patient. Consequently, the limitations of 4D-CT prevent applicability in acquiring information over timescales that represent a treatment session. MRI is highly advantageous as it is non-ionizing and provides excellent soft tissue contrast. Although real-time 3D dynamic MRI is limited by low image quality and temporal resolution, 2D dynamic MRI techniques have high fidelity and spatio-temporal resolution requisite for real-time tracking of the moving target. Furthermore, a respiration-correlated 4D-MRI can be reconstructed from multi-slice 2D dynamic MR images, enabling volumetric image processing and analysis. Therefore, 4D-MRI is an attractive solution to address breathing motion and tumor tracking obstacles in radiotherapy.

The main goal of this research is to characterize patient-specific respiration-induced tumor and surrogate motion to evaluate the accuracy and effectiveness of the surrogate-based motion management strategies currently used in clinics. Specifically, the investigators hypothesize that dynamic MRI obtained over a temporal duration consistent with radiotherapy treatments will provide spatio-temporal information of both the tumor and surrogate, and therefore can serve as a means to assess the quality of the tumor motion tracking with the surrogate. To test their hypothesis, the investigators specifically propose to 1) track and characterize the tumor and surrogate motion with 4D-MRI and 2) evaluate surrogate-based motion tracking in a cohort of patients with thoracic tumors.

External and internal surrogate-based strategies commonly used in clinics have not been appropriately validated. With the increasing adaptation of these surrogate methods for motion management, the proposed research addresses these urgent issues in clinical radiotherapy while providing a means to achieve patient-specific motion management.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed primary lung cancer (non-small cell OR small cell)
* Plan to undergo external radiation treatment of lung cancer

Exclusion Criteria:

* Patients who cannot undergo MRIs.
* Patients who have a cardiac device or other electronic or metal implant

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cancer being treated with radiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2013-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Tumor motion characterization during radiation therapy | 1 year
  To characterize patient-specific respiration-induced tumor and surrogate motion to evaluate the accuracy and effectiveness of the surrogate-based motion management strategies currently used in radiotherapy.

SECONDARY OUTCOMES:
Correlation of tumor and surrogate motion | 1 year
  Tumor and surrogate motion will be quantified by measuring the displacements from their end-exhale positions. Since the tumor may deform during motion, we will not only consider the trajectories of the center of mass but also the tumor borders. The tumor position as a function of the surrogate position will be analyzed along each moving direction. Pearson correlation coefficients and the sum of squared residual errors based on a regression analysis will be computed to provide a quantitative measure of the correlation between the surrogate and tumor positions. To measure the tumor deformation, correlations of the motion between the SI borders, AP borders, LR borders will also be computed. Although lung tumor likely does not significantly deform, this analysis will be useful for tumors that may deform significantly during motion. The motion under the different breathing patterns will be analyzed separately, and compared to each other.
Sensitivity and specificity of gating | 1 year
  Respiratory gating is one predominant technique for managing respiratory motion. Gating attempts to minimize normal tissue dose by delivering radiation during a portion of the respiratory cycle where the respiratory state is typically determined from an external surrogate as an optical signal. We will use different gating boundaries, e.g. 10%, 20% of the surrogate motion range (from mean exhale to mean inhale) on each axes as commonly used in clinical practice. Sensitivity and specificity of the gating will be computed by comparing the portion of time the surrogate is below/above the gating boundary and that the tumor is below/above the gating boundary.
Pre- and intra-treatment motion variability | 1 year
  MRI scans of the patient will be acquired pre- and intra-treatment. Tumor motion variability will be computed between these two scans. We will evaluate the correlation of the target location captured at different time points by computing target volume overlap and systematic volume shift. We will also analyze the tumor position as a function of the surrogate position for both pre- and intra-treatment scans, and will investigate how well these two distributions match. To quantitatively measure the differences, we will compute various statistical similarity measures such as correlation coefficient and mutual information. We will also calculate pre-treatment margins to account for the tumor motion using the pre-treatment retrospective 4D-MRI reconstruction, and calculate the portion of treatment time the tumor moves within or outside the specified margins during the successive scans.

CONTACTS AND LOCATIONS:
Overall Officials: Russell Hales, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States